CLINICAL TRIAL: NCT00169546
Title: Randomised, Double-blind Parallel Group Study to Assess the Bronchodilative and Bronchoprotective Properties of SERETIDE DISKUS ® Inhlaer 50/100mcg Twice Daily vs. FLIXOTIDE® Inhaler 200mcg Twice Daily.
Brief Title: Study In Airway Physiology In Children SERETIDE DISKUS ® Inhlaer and FLIXOTIDE® Inhaler Are Trademarks of GSK Group of Companies.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAM40100
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Asthma; inhaled corticosteroids
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Salmeterol/fluticasone propionate; Drug: Fluticasone propionate

INTERVENTIONS:
Drug: Salmeterol/fluticasone propionate
Drug: Fluticasone propionate
  Other Names: Salmeterol/fluticasone propionate

SUMMARY:
Comparison of two asthma treatments by lung function measures.

ELIGIBILITY:
Inclusion criteria:

* Currently receiving 200-800mcg/day beclomethasone dipropionate.
* sRAW value of 1.3 kPa's.

Exclusion Criteria:

* 3 or more courses of oral steroids in last 12 months.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2003-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
sRAW (k.Pa.s) measured before the study medication dose at the end of treatment (week 6)

SECONDARY OUTCOMES:
sRAW measured pre-dose at Week 3. sRAW measured 48 hours after last study medication dose. % symptom-free days over Weeks 1-6. % symptom-free nights over Weeks 1-6. Type and frequency of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Wellington, New Zealand
- GSK Investigational Site, Manchester, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: SAM40100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SAM40100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SAM40100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SAM40100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SAM40100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SAM40100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SAM40100 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register